CLINICAL TRIAL: NCT01418794
Title: Efficacy and Safety of the YUKON Drug Eluting Stent in Diffuse Coronary Artery Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Yaling Han, M.D. PhD, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYNH-20101010
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2010-10

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute Coronary Syndromes; Drug eluting stent; Diffused lesion
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose rapamycin group (Active Comparator): Concentration of rapamycin was 1.5%
  Interventions: Device: Low dose rapamycin stent
- High dose rapamycin group (Experimental): Concentration of rapamycin is 2.5%
  Interventions: Device: High dose rapamycin stent

INTERVENTIONS:
Device: High dose rapamycin stent — Concentration of rapamycin is 2.5%
  Arms: High dose rapamycin group
Device: Low dose rapamycin stent — Concentration of rapamycin is 1.5%
  Arms: Low dose rapamycin group

SUMMARY:
Polymer carried by drug-eluting stents may increase inflammatory response and thrombosis. Our previous study showed that polymer-free rapamycin-coated stents brings dose-dependent reduction in restenosis. This prospective, multicenter, randomized controlled clinical trials aimed to explore efficacy and safety of the YUKON drug eluting stent in diffuse coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18-85 years old, male or nonpregnant women
* asymptomatic ischemia, stable or unstable angina, old myocardial infarction patients
* at least one target lesion length ≥ 20 mm (Visual method)
* Target lesion diameter 2.5mm-4.0 mm (Visual method)
* Target lesion diameter stenosis ≥ 70%
* Patients who has indications for coronary artery bypass graft (CABG) surgery
* Patients who is voluntary, understand the purpose of the study, willing to accept angiography and clinical follow-up

Exclusion Criteria:

* Acute myocardial infarction for less than 1 week
* Bridge vascular disease
* In-stent restenosis lesions
* Patient with bleeding tendency, history of active peptic ulcer, History of cerebral hemorrhage or subarachnoid hemorrhage, history of stroke within half year, contraindications to anticoagulant therapy and antiplatelet
* Allergic to aspirin, clopidogrel or ticlopidine, heparin, contrast agent, rapamycin and metal
* Life expectancy is less than 12 months
* Patient who has participated in other clinical trials but does not meet the deadline of the primary endpoint
* Poor patient compliance
* Heart transplant recipient
* Patient who had other stent implanted within 1 year
* Patient who has multi-vessel disease(Long lesions) and has already received other stent implantation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
270-day(+60 days) in-stent late lumen loss(LLL) measured by quantitative coronary angiography (QCA) | 270 days

SECONDARY OUTCOMES:
Restenosis rate in Stent, stent proximal edge, distal edge of stent and the lesion segment | 270 days
Composite end point of major adverse cardiac events(MACE) | 30 days, 6 months, 9 months, 1 year
  Composite end point of cardiac death, all Q-wave and non-Q wave myocardial infarction, clinical-driven target lesion revascularisation
Stent thrombosis events after PCI for 24 hours, 30 days and 1 year | 24 hours, 30 days and 1 year
  according to ARC definition
Success rate of stent implantation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Ling Han, MD, Principal Investigator — Shenyang Northern Hospital
Locations (4):
- China (4):
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Shenyang Northern Hospital, Shenyang, Liaoning
  - Armed Police Force Medical College Hospital, Tianjin, Tianjin Municipality